CLINICAL TRIAL: NCT05536791
Title: Safety of Dabigatran Etexilate (DE) for Treatment of Venous Thromboembolism (VTE) and Prevention of Recurrent VTE in Paediatric Patients From Birth to Less Than 2 Years of Age: a Prospective European Non-interventional Cohort Study Based on New Data Collection
Brief Title: A Study in Europe Based on Medical Records That Looks at the Safety of Dabigatran in Children Below 2 Years of Age Who Have Had a Blood Clot and Are at Risk of Developing Another Blood Clot
Acronym: DaPaR
Status: Withdrawn | Type: Observational
Why Stopped: No patients were screened in the study.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0307
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients eligible for Dabigatran Etexilate (DE) VTE treatment and secondary VTE prevention
  Interventions: Drug: Dabigatran Etexilate (DE)

INTERVENTIONS:
Drug: Dabigatran Etexilate (DE) — Dabigatran Etexilate (DE)
  Other Names: Pradaxa®

SUMMARY:
The study is designed to collect and evaluate Dabigatran Etexilate (DE) safety in the context of routine anticoagulation care provided in the European Union (EU)/European Economic Area (EEA) for children under 2 years of age.

The non-interventional study will be conducted in paediatric hospitals or paediatric departments of EEA member states where Venous thromboembolism (VTE) patients of the evaluated age group are treated.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent from parents/care givers
* Children from birth to less than 2 years of age
* Initiation of Dabigatran Etexilate (DE) administration:

  * for treatment of Venous thromboembolism (VTE) or/and
  * prevention of recurrent VTE due to presence of unresolved clinical VTE risk factor(s).

Exclusion criteria:

* Participation in any Randomised Clinical Trial or use of any investigational product
* Any contraindications to DE according to the EU Summary of Product Characteristics (SmPC)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric patients from birth to < 2 years of age considered by investigator after screening as eligible for Dabigatran Etexilate (DE) treatment of acute Venous thromboembolism (VTE) or secondary prevention of recurrent VTE will be enrolled in the Post-Authorization Safety Study (PASS).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of any bleeding events defined as Major Bleeding Events (MBE) or Non-Major Bleeding Events (Non-MBE) | up to 6 months
  Major bleeding defined as:
  * Fatal Bleeding,
  * Clinically overt bleeding associated with a decrease in haemoglobin of at least 2 g/dL (20 g/L) in a 24-hour period,
  * Bleeding that is retroperitoneal, pulmonary, intracranial, or otherwise involves the central nervous system,
  * Bleeding that requires surgical intervention in an operating suite.
  Non-Major bleeding defined as:
  - Any overt or macroscopic evidence of bleeding that does not fulfil the criteria for major bleeding.
  (Criteria for differentiation of Major Bleeding Events (MBEs) and Non-MBEs by the Perinatal and Paediatric Haemostasis Subcommittee of the Scientific and Standardization Committee (SSC) of the International Society on Thrombosis and Haemostasis (ISTH).)

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | up to 6 months
Incidence of Serious Adverse Events (SAEs) | up to 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Netherlands (2):
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Materno Infantil Gregorio Marañón, Madrid
- Karolinska Universitetssjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com